CLINICAL TRIAL: NCT03509532
Title: A POST MARKET REGISTRY OF ABLUMINUS® SIROLIMUS ELUTING CORONARY STENT SYSTEM FOR PERCUTANEOUS INTERVENTION IN PATIENTS WITH DIABETES MELLITUS
Brief Title: DRUG ELUTING STENT FOR DIABETIC PATIENTS IN CORONARY ARTERY DISEASE TREATMENT
Acronym: DEDICATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Luca Testa, MD; PhD, IRCCS Policlinico S. Donato
Other Study IDs: DEDICATE
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PCI — PCI

SUMMARY:
Study Title A post market registry of Abluminus® sirolimus eluting coronary stent system for percutaneous intervention in patients with diabetes mellitus Purpose The purpose of this registry is to prospectively capture clinical data of ABLUMINUS® sirolimus eluting stent in patients with Diabetes Mellitus.

Investigational Device ABLUMINUS® sirolimus eluting stent consists of four components; a bare metal stent (BMS), a delivery system, the bio absorbable polymer delivery matrix and Abluminal surface coating on stent and parts of balloon in Pre-crimped condition the anti-proliferative drug, Sirolimus.

Study Design Prospective, Observational, Multi-center registry Estimated Enrolment 1000 patients

End points Primary Endpoints:

Target Lesion Failure that is composite of cardiac death, target-vessel myocardial infarction, and clinically indicated target lesion revascularisation within 12 months.

Components of the primary end point are defined as follows:

* Cardiac Death: any death due to immediate cardiac cause, deaths related to the procedure, unwitnessed death, and death of unknown cause.
* Target Vessel Myocardial infarction: categorised according to the Minnesota electrocardiographic criteria (Q-wave and non-Q-wave). Spontaneous myocardial infarction was defined as a typical rise and fall of creatinine kinase-MB fraction or troponin in the presence of at least one of several conditions: ischaemic symptoms, new pathological Q waves, ischaemic electrocardiographic changes, or pathological evidence of acute myocardial infarction. Peri-procedural myocardial infarction was defined as an increase in creatinine kinase to more than twice the normal value with increased values of confirmatory biomarkers (creatinine kinase-MB fraction or troponin higher than usual). Target-vessel-related myocardial infarction was one related to the target vessel or that could not be clearly related to another vessel.
* Target Lesion Revascularisation: any repeat percutaneous or surgical intervention due to a stenosis or occlusion within the device of the index procedure.

Secondary Endpoints

* Stent thrombosis [Time Frame: 1 month, 12 months, yearly]. Definite and probable stent thrombosis according to ARC definitions;
* Cardiac death [Time Frame: 1 month, 12 months, yearly]
* Target Vessel Myocardial infarction [Time Frame: 1 month, 12 months, yearly]
* Target Lesion Revascularisation [Time Frame: 1 month, 12 months, yearly]
* Device Success at 24 hours
* Lesion Success at 24 hours
* Procedural Success at 24 hours Eligibility Eligible Age: 18 Years and older. Eligible Genders: Both. Inclusion Criteria
* The patient must be at least 18 years of age.
* Diabetic patient having clinical evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia or positive functional study; acute coronary syndromes will be considered).
* The patient is an acceptable candidate for percutaneous trans-luminal coronary angioplasty (PTCA) stenting and emergent coronary artery bypass graft (CABG) surgery.
* Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation (no limitation on the number of treated lesions, vessel and lesion length);
* Patients included are those for whom the physician has already considered worthwhile the use of Abluminus Stent according to the indications provided by the IFU;
* Patient provides written informed consent;
* Patient agrees to all required follow-up procedures and visits. Exclusion Criteria • The patient has a known hypersensitivity or contraindication to any of the following medications:Heparin, Aspirin, Both Clopidogrel and TIclopidine, Sirolimus, paclitaxel, ABT 578Stainless steel, Cobalt, biodegradable PLLA polymer.
* Patients with hypersensitivity to contrast media who cannot be treated with adequate prophylaxis.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrolment into this study.
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
* Previous coronary intervention on target vessel.
* Non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Lesions not allowing a complete balloon inflation or stent deployment. Clinical Follow up At Discharge, 1 month, 6 months, 12 months, yearly.

DETAILED DESCRIPTION:
DEDICATE Registry:

DRUG ELUTING STENT FOR DIABETIC PATIENTS IN CORONARY ARTERY DISEASE TREATMENT

A POST MARKET REGISTRY OF ABLUMINUS® SIROLIMUS ELUTING CORONARY STENT SYSTEM FOR PERCUTANEOUS INTERVENTION IN PATIENTS WITH DIABETES MELLITUS

Version 1.0

Principal Investigator Dr. Luca Testa, MD, PhD Head of Coronary Revascularization Unit Head of Clinical Research Unit Department of Cardiology, IRCCS Policlinico S. Donato, San Donato M.ne, Milan, Italy Email: luctes@gmail.com

Chairperson Dr. Francesco Bedogni, MD Head of Cardiology IRCCS Policlinico S. Donato, San Donato M.ne, Milan, Italy

Protocol Signature Page

Principal Investigator (Coordinator Center)

Investigate site IRCCS Policlinico San Donato

Name Dr. Luca Testa

Signature ______________________

Date _____________________

Chairperson (Coordinator Center)

Investigate site IRCCS Policlinico San Donato

Name Dr. Francesco Bedogni

Signature ______________________

Date _____________________

Principal Investigator

Investigate site ___________________

Name __________________

Signature ______________________

Date _____________________

Protocol summary

Study Title A post market registry of Abluminus® sirolimus eluting coronary stent system for percutaneous intervention in patients with diabetes mellitus Purpose The purpose of this registry is to prospectively capture clinical data of ABLUMINUS® sirolimus eluting stent in patients with Diabetes Mellitus.

Investigational Device ABLUMINUS® sirolimus eluting stent consists of four components; a bare metal stent (BMS), a delivery system, the bio absorbable polymer delivery matrix and Abluminal surface coating on stent and parts of balloon in Pre-crimped condition the anti-proliferative drug, Sirolimus.

Study Design Prospective, Observational, Multi-center registry Estimated Enrolment 1000 patients

End points Primary Endpoints:

Target Lesion Failure that is composite of cardiac death, target-vessel myocardial infarction, and clinically indicated target lesion revascularisation within 12 months.

Components of the primary end point are defined as follows:

* Cardiac Death: any death due to immediate cardiac cause, deaths related to the procedure, unwitnessed death, and death of unknown cause.
* Target Vessel Myocardial infarction: categorised according to the Minnesota electrocardiographic criteria (Q-wave and non-Q-wave). Spontaneous myocardial infarction was defined as a typical rise and fall of creatinine kinase-MB fraction or troponin in the presence of at least one of several conditions: ischaemic symptoms, new pathological Q waves, ischaemic electrocardiographic changes, or pathological evidence of acute myocardial infarction. Peri-procedural myocardial infarction was defined as an increase in creatinine kinase to more than twice the normal value with increased values of confirmatory biomarkers (creatinine kinase-MB fraction or troponin higher than usual). Target-vessel-related myocardial infarction was one related to the target vessel or that could not be clearly related to another vessel.
* Target Lesion Revascularisation: any repeat percutaneous or surgical intervention due to a stenosis or occlusion within the device of the index procedure.

Secondary Endpoints

* Stent thrombosis [Time Frame: 1 month, 12 months, yearly]. Definite and probable stent thrombosis according to ARC definitions;
* Cardiac death [Time Frame: 1 month, 12 months, yearly]
* Target Vessel Myocardial infarction [Time Frame: 1 month, 12 months, yearly]
* Target Lesion Revascularisation [Time Frame: 1 month, 12 months, yearly]
* Device Success at 24 hours
* Lesion Success at 24 hours
* Procedural Success at 24 hours Eligibility Eligible Age: 18 Years and older. Eligible Genders: Both. Inclusion Criteria
* The patient must be at least 18 years of age.
* Diabetic patient having clinical evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia or positive functional study; acute coronary syndromes will be considered).
* The patient is an acceptable candidate for percutaneous trans-luminal coronary angioplasty (PTCA) stenting and emergent coronary artery bypass graft (CABG) surgery.
* Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation (no limitation on the number of treated lesions, vessel and lesion length);
* Patients included are those for whom the physician has already considered worthwhile the use of Abluminus Stent according to the indications provided by the IFU;
* Patient provides written informed consent;
* Patient agrees to all required follow-up procedures and visits. Exclusion Criteria • The patient has a known hypersensitivity or contraindication to any of the following medications:Heparin, Aspirin, Both Clopidogrel and TIclopidine, Sirolimus, paclitaxel, ABT 578Stainless steel, Cobalt, biodegradable PLLA polymer.
* Patients with hypersensitivity to contrast media who cannot be treated with adequate prophylaxis.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrolment into this study.
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
* Previous coronary intervention on target vessel.
* Non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Lesions not allowing a complete balloon inflation or stent deployment. Clinical Follow up At Discharge, 1 month, 6 months, 12 months, yearly.

CONTENTS

1. BACKGROUND AND INTRODUCTION 7
2. RISK ANALYSIS 9
3. AIM OF THE REGISTRY 11
4. REGISTRY DESIGN 11
5. ENDPOINT 11
6. REGISTRY POPULATION 12
7. REGISTRY PROCEDURES 13
8. ANTITHROMBOTIC TREATMENT 14
9. FOLLOW-UP PERIOD 15
10. SERIOUS ADVERSE EVENT REPORTING 15
11. MACE ADJUDICATION 16
12. STATISTICAL ANALYSIS 16
13. QUALITY CONTROL AND ASSURANCE 16
14. ETHICAL CONSIDERATION 17

<!-- -->

1. BACKGROUND AND INTRODUCTION

   Era of Percutaneous Coronary Intervention (PCI) started with plain old balloon angioplasty (POBA) and progressed to bare metal stent (BMS) and then to drug-eluting stent (DES). In DES, polymer was used in addition to the drug, so that it could hold the drug on the stent platform and could facilitate controlled drug release. Thus, drug and polymer became hallmark of DES [1].

   Current DES consist of a metal stent platform and a therapeutic agent, which is either directly immobilized on the stent surface or released from a polymer matrix. While drug-eluting stents without surface polymer are available, the reduction in angiographic and clinical restenosis is less potent and appears therefore less promising for clinical utilization. In contrast, polymer-based, drug-eluting stents allow for controlled release of therapeutic agents at the site of injury [2].

   The most effective drugs utilized with drug-eluting stents for prevention of restenosis up to this point in time have been Sirolimus and Paclitaxel. Both drugs are highly lipophilic and show rapid and strong uptake in arterial wall tissue. In addition, Sirolimus and paclitaxel have been shown to reduce smooth muscle cell proliferation and neo-intimal hyperplasia, the principal cause of restenosis after coronary stenting in experimental models. Sirolimus and Paclitaxel have the same effect on cells proliferation, but with a different mode of action.A recent meta-analysis of drug-eluting stent trials confirmed the reduction in restenosis and repeat revascularization procedures for polymer-based, drug-eluting stents. Moreover, the rates of death and myocardial infarction were comparable to those with bare-metal stents, attesting to the safety of these devices, which have been approved by the US Food and Drug Administration.

   Patients with diabetes mellitus referred for percutaneous coronary intervention (PCI) represent one of the greatest challenges for the interventional cardiologist. Restenosis continues to be the major limitation of PCI, particularly in patients with diabetes [2]. Restenosis rates after balloon angioplasty in diabetic patients can be very high (up to 63%), and although stenting has been shown to decrease these rates, diabetic patients continue to have significantly higher restenosis rates and clinical events following PCI. Slight elevations in fasting blood glucose levels, the need for insulin, and suboptimal blood glucose control may have a significant impact on the prognosis. Drug-eluting stents (DES) have been shown to have a considerably lower risk of restenosis and as a result, there is growing interest in using such stents to treat coronary lesions in complex scenarios. Sub studies carried out in diabetic patients from large clinical trials conducted with DES have found considerable decreases in the risk of restenosis and new revascularizations. [3,4] Nevertheless, despite the availability use of DES, diabetic patients show a higher risk than non-diabetics.Hyperinsulinemia and insulin resistance are implicated in a variety of molecular mechanisms that could predispose diabetics to a higher incidence of restenosis.

   The purpose of this registry is to capture clinical data of ABLUMINUS® sirolimus eluting stent in in real world, all come patients with Diabetes Mellitus.

   1.1 Device Description

   The device ABLUMINUS® Sirolimus eluting coronary stent integrates well known and accepted Sirolimus drug on the proven CYGNUS Cobalt chromium platform with biodegradable polymer matrix.

   The device ABLUMINUS® sirolimus eluting stent system has a combination of inactive and active component. The active component is Sirolimus drug. The inactive component is PLLA polymer (biodegradable polymer). The polymer-drug combination is applied solely to a unique abluminal coating technology known as "ënvisõlution™ Technology" which is a highly effective drug delivery technology with target specific coating in abluminal configuration on stent and parts of balloon. It also uses biodegradable polymer to achieve longer drug release.

   The stent platform is a thin strut (73 microns) of L605cobalt chromium stent with open and closed cell (hybrid) design, which provides good radial strength and side branch accessibility. The thin struts enhance the trackability and gives lower crossing profile to the device for navigating through difficult and tortuous lesions. The delivery system is a Rapid exchange (Rx) System.

   It is expected that ABLUMINUS® sirolimus eluting stent system will significantly reduce delay in healing and thrombosis events, while providing comparable results, regarding restenosis, to other DES systems on the market.

   1.2 Therapeutic Agent-Sirolimus Drug

   Sirolimus is a cytostatic drug used for treatment of various disease in Humans. The drug works on FKBP-12 protein and inhibits growth factor-simulated cell proliferation. Sirolimus forms a complex with FKBP Protein that inhibits the cell cycle between G0 and G1 phase. This results in interruption of the cascade governing cell growth, metabolism and proliferation.

   1.3 STENT PLATFORM ABLUMINUS® sirolimus eluting stent system is a combination product comprised of two key components: the Stent (which includes the active pharmaceutical ingredient (API) Sirolimus drug incorporated into a bio-degradable polymer coating), and delivery catheter. A balloon expandable L605 chromium cobalt stent with bio-degradable polymer coating containing Sirolimus drug is pre-mounted onto a highly deliverable semi-compliant rapid exchange delivery system. The delivery catheter has two radiopaque markers, which mark the ends of the stent to facilitate proper positioning and placement. The catheter has hydrophilic coating facilitating easy delivery of the system.

   The Stent has a biodegradable polymer matrix consisting of Poly L Lactic acid (PLLA) which has been wide spread application in medical devices. The Poly lactic acid, its co-polymers and mixtures have been evaluated in pre-clinical studies and clinical studies around the world, revealing favourable bio-compatibility profile. The bio-degradable polymer has been demonstrated to be safe when used as an implant or drug release-control polymer for both animal and humans.
2. RISK ANALYSIS

   As with any patient undergoing percutaneous coronary intervention, subject in this registry may experience adverse events and/or outcomes that may include, but are not necessarily limited to the following:
   * Abrupt stent closure or failure to expand the stent
   * Abrupt vessel closure or spasm
   * Acute myocardial infarction
   * Allergic reaction to anti-coagulation and/or anti thrombotic therapy, contrast material, or stent and/or delivery system materials
   * Aneurysm, pseudo aneurysm or arteriovenous fistula
   * Arrhythmias, including ventricular fibrillation and ventricular tachycardia
   * Cardiac tamponade
   * Cardiogenic shock
   * Death
   * Dissection, perforation, or rupture of the coronary artery
   * Emboli, distal (air, tissue or thrombic emboli)
   * Emergency coronary artery bypass graft (CABG) as a result of damage to the stent / injury to the vessel
   * Fever
   * Hematoma at insertion site
   * Haemorrhage requiring transfusion
   * Hypotension/hypertension
   * Infection and/or pain at site of insertion
   * Late stent thrombosis/ stent thrombosis/ occlusion
   * Perforation or rupture of artery
   * Peripheral ischemia or peripheral nerve injury
   * Stroke or transient ischemia attack
   * Renal failure
   * Restenosis of stented segment
   * Stent migration or stent embolization
   * Total occlusion of coronary artery
   * Unstable angina

   Adverse events that may be associated with Sirolimus drug coating:
   * Allergic/immunologic reaction to drug or stent coating
   * Alopecia
   * Anaemia
   * Blood product transfusion
   * Gastrointestinal symptoms
   * Haematologicaldyscrasia (including leukopenia, neutropenia, thrombocytopenia)
   * Hepatic enzyme changes
   * Histological changes in vessel wall, including inflammation, cellular damage or necrosis
   * Myalgia/Arthralgia
   * Peripheral neuropathy

   Appropriate contraindications and warnings are also included in the instructions for use provided with the device. Interventional cardiologists are invited to participate as investigators in this registry. All clinicians will have experience with the treatment and control procedures and have been trained on the use / implantation of a Drug Eluting stent system.
3. AIM OF THE REGISTRY

   The purpose of this registry is to capture clinical data of ABLUMINUS® sirolimus eluting stent in real world, all comer patients with Diabetes Mellitus.
4. REGISTRY DESIGN

   Prospective, Observational, Multi-center clinical registry to be conducted in Italy at 15 Interventional cardiology centers. 1000 patients will be enrolled and evaluated. All the patients will be followed up for up to 5 years.

   4.1 Treatment Strategy

   The investigator will determine the treatment strategy. It is recommended that each enrolling investigator review the most recent IFU to assess contraindications, warnings, and precautions for treating potential patients.
5. ENDPOINT

   5.1 Primary endpoints

   Target Lesion Failure, which is composite of cardiac death, target-vessel myocardial infarction, and clinically indicated target lesion revascularisation within 12 months.

   Components of the primary end point are defined as follows:

   • Cardiac Death: any death due to immediate cardiac cause, deaths related to the procedure, unwitnessed death, and death of unknown cause.
   * Target Vessel Myocardial infarction: categorized according to the Minnesota electrocardiographic criteria (Q-wave and non-Q-wave). Spontaneous myocardial infarction was defined as a typical rise and fall of creatinine kinase-MB fraction or troponin in the presence of at least one of several conditions: ischemic symptoms, new pathological Q waves, ischemic electrocardiographic changes, or pathological evidence of acute myocardial infarction. Peri-procedural myocardial infarction was defined as an increase in creatinine kinase to more than twice the normal value with increased values of confirmatory biomarkers (creatinine kinase-MB fraction or troponin higher than usual). Target-vessel-related myocardial infarction was one related to the target vessel or that could not be clearly related to another vessel.
   * Clinically indicated target lesion revascularisation: any repeat percutaneous or surgical intervention due to a stenosis or occlusion within the device of the index procedure 5.2 Secondary endpoints
   * Stent thrombosis [Time Frame: 1 month, 12 months, yearly]: Definite and probable stent thrombosis according to ARC definitions.
   * Cardiac death [Time Frame: 1 month, 12 months, yearly]
   * Target Vessel Myocardial infarction [Time Frame: 1 month, 12 months, yearly]
   * Target Lesion Revascularisation [Time Frame: 1 month, 12 months, yearly]
   * Device Success at 24 hours
   * Lesion Success at 24 hours
   * Procedural Success at 24 hours
6. REGISTRY POPULATION

6.1 Number of patients 1000 patients will be enrolled at 15 interventional cardiology sites in Italy. Duration of enrollment will be 12 months.

6.2 Type of Patient Patients eligible for PCI (Percutaneous Coronary Intervention) with lesions suitable for stent implantation and having diabetes Mellitus will be included according to the inclusion and exclusion criteria specified below. The inclusion criteria will be kept comprehensive to reflect routine clinical practice of treatment (Real world Scenario-All comer patients).

1. Inclusion Criteria

   1. The patient must be at least 18 years of age. 2. Diabetic patient having clinical evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia or positive functional study; acute coronary syndromes will be considered).

   3. The patient is an acceptable candidate for percutaneous trans luminal coronary angioplasty (PTCA),stenting and emergent coronary artery bypass graft (CABG) surgery.

   4. Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation (no limitation on the number of treated lesions, vessel and lesion length); 5. Patients included are those for whom the physician has already considered worthwhile the use of Abluminus Stent according to the indications provided by the IFU; 6. Patient provides written informed consent; 7. Patient agrees to all required follow-up procedures and visits.
2. Exclusion Criteria

   1. The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Both Clopidogrel and Ticlopidine, Sirolimus, Paclitaxel, ABT 578 Stainless steel, Chromium; Cobalt, biodegradable PLLA polymer.
   2. Patients with hypersensitivity to contrast media who cannot be treated with adequate prophylaxis
   3. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study;
   4. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions;
   5. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
   6. Previous coronary intervention on target vessel;
   7. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment);
   8. Lesions not allowing a complete balloon inflation or stent deployment.

   7. REGISTRY PROCEDURES

   7.1 Patient Information

   Eligible patients will be informed about the registry and have to sign informed consent before or after the procedure (see Appendix I: informed consent form).

   7.2 Baseline Evaluation

   At inclusion into registry, the following routine examination, if performed, will be captured:

   1. Physical examination and relevant medical history; 2. Angina status; 3. Routine laboratory tests including complete blood count (CBC), blood chemistry, blood sugar and lipids, CK and/or CK-MB prior to the procedure. In case of acute myocardial infarction or infarct extension we suggest CK and/or CK-MB immediately prior to the procedure and serial measurements every 8 hours after the procedure until the peak CK level has been defined 4. 12-lead electrocardiogram before the procedure.

   7.3 Stent Implantation

   During the index procedure, only ABLUMINUS® sirolimus eluting stent system will be implanted. Using the instruction for use (IFU), provided with the device, the investigator will choose the appropriate length and diameter of the stents to be implanted by visual estimation.

   The choice of the length of the stent should ensure complete coverage of the lesion. If more than one stent is implanted, at least 2 mm overlap should be achieved. In case of insufficient stent expansion, the stent will be post-dilated with an appropriately sized balloon.

   Treatment of multiple target vessels (within the same procedure) and staged procedures which occur within 90 days of the initial implant procedure are allowed. ABLUMINUS® sirolimus eluting stent system implanted in non-target vessels after > 90 days after the initial implant procedure will not be followed under the ABLUMINUS® sirolimus eluting stent system registry protocol.

   As such, any subsequent treatment of the lesion already present at the time of baseline procedure will be considered as a staged procedure, instead of a repeat PCI. In the CRF (Case Report Form), the investigator will complete a 'staged procedure' module indicating that this lesion was present at the time of first procedure. The lesions diagnosed and treated at the later stages will not be considered as "repeat" revascularization.

   For each individual lesion treated, a separate lesion form in the CRF needs to be completed. Every vessel in which anABLUMINUS® sirolimus eluting stent system is implanted (or in which an attempt to implant anABLUMINUS® sirolimus eluting stent system is made) within 90 days of the initial implant procedure is considered a target vessel.

   For patient undergoing a staged procedure, the follow up schedule will be calculated from the date of initial ABLUMINUS® sirolimus eluting stent system implant procedure.

   8. ANTITHROMBOTIC TREATMENT

   Pre- procedure*: Aspirin 75mg minimum;

   Patients without any therapy: clopidogrel bisulphate: loading dose of 300-600mg per os before or during the procedure;

   Patient on clopidogrel therapy (within 7 days prior) no loading dose required.

   Ticagrelor or Prasugrel in the case of Acute Coronary Syndromes

   During Procedure*: At least 5000IE or 70-100IE/Kg unfractioned heparin to maintain an ACT > 250 seconds during the procedure.**

   Post-procedure*: DAPT Therapy for at least 6 months (IFU), or longer according to current Guidelines Aspirin 75mg per os life long.

   *Or according to standard clinical practice. / **The use of GP IIB/ IIIA inhibitors is left to the discretion of the operator.

   9. FOLLOW-UP PERIOD

   Patients will be followed after hospital discharge up to 5 years after the index procedure. This includes telephone contacts to obtain information regarding medical history, cardiovascular drug use, hospitalizations, and adverse events at 1 month, 6 months 12 months, and then yearly post procedure. Apart from clinical follow -ups there is angiographic follow-up which is clinically driven (symptom driven).

   10. SERIOUS ADVERSE EVENT REPORTING

   10.1 Serious Adverse Events (SAEs)

   An adverse event (AE) is report as serious which lead to:
   * Death
   * Life-threatening illness or injury, or
   * Permanent impairment of a body structure or a body function, or
   * In-patient or prolonged hospitalization (see note below), or
   * Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.

   Note: For the purposes of this study, in-patient hospitalization is defined as the subject being admitted to the hospital, with the exception of any planned hospitalization for a pre-existing condition or a procedure required by the local standard of care, which do not have to be reported as an SAE.

   All serious adverse events must be reported to the Principal Investigator within 24 hours of discovery or notification of the event and to the local EC, as per local requirements.

   The Principal Investigator is responsible for reporting adequate information on SAEs that may be related to the study device to the regulatory authorities per country's applicable reporting requirements.

   10.2 Unanticipated Serious Adverse Device Effect (USADE)

   Any serious adverse effect on the health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

   Unanticipated Adverse Device Effects must be reported to the manufacturer as soon as possible following the standard vigilance route. Reporting the event ONLY in the CRF is not an option.

   11. MACE ADJUDICATION

   All registry devices related Major Adverse Cardiac Events (MACE) will be reviewed & classified by the treating physician. In case of a stent thrombosis or severe stent restenosis, these events will verify the stent thrombosis & determine the % Diameter Stenosis (DS) by QCA.

   12. STATISTICAL ANALYSIS

   12.1 Analysis Population All patients who are successfully registered will be included in the analysis.

   12.2 Sample Size Calculations and Assumptions Being this an observational registry aiming at quantifying effect estimates without direct comparisons to literature benchmarks, we proceeded without a formal power analysis. As the main analysis is a pooled analysis of all included patients, an overall and comprehensive analysis is planned as the primary analytical approach to reflect real-world patients and practice.

   12.3 Statistical Analyses Continuous endpoints will be summarized by presenting the total number of patients, mean, standard deviation, median, minimum, and maximum. Tabulation of categorical parameters will include counts and percentages. Survival analysis will be performed with the Kaplan-Meier method. Statistical inference will be based on the computation of 95% confidence intervals using the adjusted Wald method. Additional analyses will involve key subgroups defined according to baseline and procedural features, with statistical significance set at the 5% 2-tailed level. Specifically, Student t, Fisher exact, and log-rank tests will be used for such bivariate analyses, whereas multivariable linear regression, logistic regression, and Cox proportional hazard analyses will be used to adjust for confounders.

   13. QUALITY CONTROL AND ASSURANCE

   13.1 Quality Assurance The Principal Investigator of the Centre is responsible for the overall clinical management of patients admitted to his center, and assumes global responsibilities for him and his staff and the data obtained from study participants; he ensures compliance with the protocol, laws and regulations, ensures informed consent to be signed and that the CRF is accurate and complete.

   In accordance with Italian law and the ICH/GCP guidelines, the investigators and the institution will allow representatives of regulatory agencies and Ethics Committee direct access for review of the original documentation of patients, to verify compliance with the procedures and the veracity of the data.

   13.2 Source Data The investigator assures that medical files are appropriately stored and completed. Each follow up contact will be reported in the source data & should at least contain the information collected by the registry. The investigator assures that medical files and case record forms are accessible for inspection by Competent Authorities.

   13.3 Monitoring The study will be performed according to "good clinical practice ". The collection of personal, procedural and clinical data of patients must take place into the electronic CRF, to which will only have access the individual investigators and the study principal investigator (Dr Luca Testa) as "administrator ".

   13.4 Publication policy All study investigators are committed to publishing the results at both conferences and international journals. The P.I. of the study will have the right to present the main results before other investigators and will be the owner of the data. After obtaining the consent of the P.I., the other experimenters will publish and present the full or partial results of the study.

   All investigators undertake to publish the study results, whether they are positive, negative, or unexpected.

   14 ETHICAL CONSIDERATION

   14.1 General Guidelines This registry will be conducted in accordance with ICH- GCP (Good Clinical Practices). The registry will be performed in accordance with the Declaration of Helsinki and ISO 14155:2011 and MED DEV 2.7.1 rev. 3.

   14.2 Ethics Committee The protocol, informed consent form and other registry-related documents will be submitted to the Institutional or Local Ethics Committee, if applicable or are required for approval to initiate.

   14.3 Informed Consent A signed Informed Consent (sample attached) must be obtained before enrolment. Importantly, patients' participation in the study is voluntary, thus, they may decide to terminate their involvement at any time by withdrawing consent.

   Bibliography

   1) Stefanini GG, Holmes DR Jr. Drug-eluting coronary-artery stents. N Engl J Med 2013;368:254-65.

   2) Serruys PW, H.E. Luijten, K.J. Beatt, et al. Incidence of restenosis after successful coronary angioplasty: a time-related phenomenon. A quantitative angiographic study in 342 consecutive patients at 1, 2, 3, and 4 months, Circulation 1988;77(2):361-371.

   3) Fihn SD, Blankenship JC, Alexander KP, et al. 2014 ACC/AHA/AATS/PCNA/SCAI/STS focused update of the guideline for the diagnosis and management of patients with stable ischemic heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines, and the American Association for Thoracic Surgery, Preventive Cardiovascular Nurses Association, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol 2014; 64:1929-49.

   4) Windecker S, Kolh P, Alfonso F, et al. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS) developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J 2014; 35:2541-619.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Diabetic patient having clinical evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia or positive functional study; acute coronary syndromes will be considered).
* The patient is an acceptable candidate for percutaneous trans-luminal coronary angioplasty (PTCA) stenting and emergent coronary artery bypass graft (CABG) surgery.
* Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for stent implantation (no limitation on the number of treated lesions, vessel and lesion length);
* Patients included are those for whom the physician has already considered worthwhile the use of Abluminus Stent according to the indications provided by the IFU;
* Patient provides written informed consent;
* Patient agrees to all required follow-up procedures and visits.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:Heparin, Aspirin, Both Clopidogrel and TIclopidine, Sirolimus, paclitaxel, ABT 578Stainless steel, Cobalt, biodegradable PLLA polymer.
* Patients with hypersensitivity to contrast media who cannot be treated with adequate prophylaxis.
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrolment into this study.
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions
* Previous coronary intervention on target vessel.
* Non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Lesions not allowing a complete balloon inflation or stent deployment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Pol. San Donato, Milan, Italy

IPD SHARING:
Plan to Share IPD: No